CLINICAL TRIAL: NCT05628506
Title: Measurement of Iodolipids in the Thyroid Gland and Other Biological Samples
Acronym: IODOLIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Gerasimos Sykiotis (Other)
Responsible Party: Sponsor-Investigator, Prof. Gerasimos Sykiotis, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IODOLIP Study
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — Potassium Iodide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Drug: Potassium iodide
- control group (No Intervention)

INTERVENTIONS:
Drug: Potassium iodide — Patients will receive a single oral administration of a pharmacological dose (97.5 mg) of potassium iodide 20±4 hours before surgery.
  Arms: intervention group

SUMMARY:
The research project is an open, parallel-group, single centre, randomized controlled trial that aims to assess the feasibility of measuring iodolipids in thyroid samples of patients during routine thyroid surgery.

DETAILED DESCRIPTION:
Twenty subjects will be included. Patients are randomized 1:1 to receive either a single oral administration of a pharmacological dose of potassium iodide 20±4 hours before surgery (10 patients), or nothing (10 patients):

* The dose administered will be 97.5 mg,
* Patients allocated to the control group will not receive any drug.

Two thyroid samples will be taken from the surgical specimen by a pathologist. Each sample will have a weight of approximatively 1 g, corresponding to a volume of approximately 1 cm3. We will select material containing tissue that corresponds to normal thyroid parenchyma (according to the preoperative ultrasound and direct inspection by the pathologist intraoperatively). The sample will be taken in the dedicated room next to the operating room by a pathologist who will confirm that the targeted area has no visible macroscopic lesion. In case of doubt, an alternative area free of lesion will be selected by the pathologist.

Patients are unblinded. The total maximum duration of the study for an individual patient is 42 days. The total duration of the clinical trial will be 3 years in order to include 20 patients.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all of the following inclusion criteria are eligible for the study:

1. Patients with the capacity for discernment and who agree to participate in the study and sign the consent.
2. Age ≥18 years.
3. Indication for thyroid surgery due to either nontoxic single thyroid nodule (WHO disease classification 5A01.1) or nontoxic multinodular goitre (WHO disease classification 5A01.2).
4. Normal thyroid function without anti-thyroid medication. This is ascertained by at least one serum TSH value within the reference range in the three months before surgery (if multiple values are available, the latest value should be normal). If no TSH values are available, a blood draw will be performed to measure TSH.

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to exclusion of the patient:

1. Women who are pregnant or breastfeeding (a urine pregnancy test will be done at Visit 2 before randomization if applicable).
2. Intention to become pregnant during the course of the study.
3. Alcohol or drug abuse within the past 6 months.
4. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the patient.
5. Participation in another study with investigational drug within the 30 days preceding and during the present study.
6. Use, within the last month before the scheduled surgery, of iodine-containing medications, i.e., iodine-containing anti-cough syrups or iodine-containing disinfectants. Non-iodine-containing anti-cough syrups and non-iodine-containing disinfectants are authorized.
7. Use, within the last month before the scheduled surgery, of iodine-containing radiological contrast media. Non-iodine-containing radiological contrast media are authorized.
8. Susceptibility to iodine-induced hyperthyroidism (i.e., toxic adenoma or toxic multinodular goiter, or previous episode of iodine-induced hyperthyroidism according to the medical history).
9. Serum TSH (thyroid-stimulating hormone) level below the lower limit of the reference range.
10. Graves' disease.
11. Susceptibility to iodine-induced hypothyroidism (history of thyroid surgery, Hashimoto's thyroiditis, history of subacute or destructive thyroiditis).
12. Titer of serum thyroid autoantibodies (anti-TSH receptor, anti-thyroperoxydase or antithyroglobulin) above the reference range.
13. History of sialadenitis, regardless of etiology.
14. History of allergic reactions (any grade) to radiological contrast media, iodine-containing disinfectants, anti-cough medications, or seafood; and known hypersensitivity to iodine.
15. History of allergic reactions (any grade) to the excipients of the ""IODURE DE POTASSIUM 65 AApot cpr 65 mg" drug: lactosum anhydricum, cellulosum microcristallinum, magnesii stearas.
16. Severe intolerance to lactose or galactose (patients having been recommended by their physician to adhere to a strict regime free of the offending agent).
17. Concurrent treatment with lithium.
18. Concurrent treatment with potassium-sparing diuretics.
19. Nodule diagnosed as thyroid carcinoma or suspicious for thyroid carcinoma based on the results of a fine-needle aspiration biopsy or a tru-cut biopsy (if performed during the routine patient work-up as per standard indications).
20. Patients with hyperkalemia.
21. Dermatitis herpetiformis.
22. Congenital myotonia.
23. Hypocomplementemic urticaria/vasculitis.
24. Chronic obstructive pulmonary disease
25. Asthma
26. Heart failure stage B, C or D
27. Impaired renal function (eGFR <60 ml/min/1.73 m2)
28. Normal urinary iodine concentration on the day of surgery (determined retrospectively).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Mean 2-iodoxehadecanal and delta-iodolactone in the thyroid sample | 20±4 hours after administration of potassium iodide